CLINICAL TRIAL: NCT02279069
Title: Comparison Between Classical 4-point Canne and 4-roll Canne on Gait Parameters (Gait Speed and Energy Cost) as Walking Aids After Stroke. A Multicentric Randomized Controled Cross-over Study
Brief Title: 4-point vs 4-roll Canne as Walking Aids After Stroke
Acronym: 4roll
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Deltombe Thierry, Professeur Clinique, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MG-4roll-53/2014
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Stroke
Keywords: stroke; walking; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4-point canne (Active Comparator): Stroke patients walk with 4-point canne
  Interventions: Device: 4-roll canne
- 4-roll canne (Experimental): Stroke patients walk with 4-roll canne
  Interventions: Device: 4-roll canne

INTERVENTIONS:
Device: 4-roll canne

SUMMARY:
Stroke patients frequently necessitate walking aids such as 4-point canne. However, the 4-point canne has to be lifted by the patient which limited gait speed. The adjunction of small wheel below the 4 point of the canne (4-roll) gives the possibility to the patient to walk without having to lift the canne as it will roll over the ground.

The aim of our study is to compare gait parameters (gait speed and energy cost) with a classical 4-point canne and with 4-roll canne.

DETAILED DESCRIPTION:
Stroke patients frequently need walking aids such as 4-point canne. However, the 4-point canne has to be lifted by the patient which limited gait speed. The adjunction of small wheel below the 4 point of the canne (4-roll) gives the possibility to the patient to walk without having to lift the canne as it will roll over the ground.

OBJECTIVE To compare the gait parameters with a 4-point canne and with a 4-roll canne METHODS The investigators will recruited stroke patients who necessitate 4 point-canne as walking aids. A 10 meters walking test, a 6 minutes walking test, an estimated energy cost and a patient's satisfaction will be monitored with a 4-point canne (day 1) and with a 4-roll canne (day 2) in a cross-over study. The first tested device will be randomized.

PERSPECTIVE The investigators hope to demonstrate that a 4-roll canne makes possible to walk faster in a safe way after stroke

ELIGIBILITY:
Inclusion Criteria:

* post stroke patient
* able to walk 10 meters

Exclusion Criteria:

* cognitive impairment limiting walking capacities
* need support when walking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
10 meters walking test at spontaneous speed | 2 days

SECONDARY OUTCOMES:
10 meters walking test at fast speed | 2 days
6 minutes walking test | 2 days
Borg scale for perceived exertion | 2 days
Visual analogic scale for personal satisfaction | 2 days
Energy cost | 2 days
  Extrapolated from heart rate while walking

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Deltombe, MD, Principal Investigator — CHU Dinant Godinne / UcL Namur; Geoffroy Dellicour, PT, Principal Investigator — Centre Neurologique William Lennox Ottignies
Locations (1):
- Deltombe Thierry, Yvoir, Belgium